CLINICAL TRIAL: NCT01185054
Title: Is Electrolyte Maintenance Solution Required in Low-Risk Children With Gastroenteritis?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000017642
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis
Keywords: Pediatrics; Gastroenteritis; Oral Rehydration; Electrolyte Maintenance Solution
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluids as Tolerated (FAT) Group (Experimental): The FAT group will receive ½ strength apple juice and will form the experimental group in this study.
  Interventions: Other: ½ strength apple juice
- Electrolyte Maintenance Solution (EMS) (Active Comparator): The EMS group will form the control group as solutions such as Pediatric Electrolyte® are routinely recommended for use in children with gastroenteritis.
  Interventions: Other: Pediatric Electrolyte

INTERVENTIONS:
Other: ½ strength apple juice — For each episode of diarrhea 10 ml/kg of fluid will be given and for each episode of vomiting 2 ml/kg will be given. If the child does not like the solution another fluid can be used.
  Arms: Fluids as Tolerated (FAT) Group
Other: Pediatric Electrolyte — For each episode of diarrhea 10 ml/kg of fluid will be given and for each episode of vomiting 2 ml/kg will be given. If the child does not like the solution another electrolyte maintenance fluid can be used. Fluids containing non-physiological concentrations of glucose and electrolytes (carbonated drinks, sweetened fruit juices, water) will be discouraged.
  Other Names: Oral Electrolyte Maintenance Solution
  Arms: Electrolyte Maintenance Solution (EMS)

SUMMARY:
The objective of this study is to clarify the current standard of care by determining if Electrolyte Maintenance Solution (EMS) is truly the optimal fluid to be used in low-risk children who present to an Emergency Department (ED) with < 72 hours of vomiting or diarrhea.

DETAILED DESCRIPTION:
Gastroenteritis remains a major cause of morbidity amongst Canadian children. The primary treatment focus revolves around the use of Oral Rehydration Therapy (ORT) to treat dehydration and replace intravascular volume. Since diarrheal disease in Canadian children usually results in mild dehydration and minimal sodium losses, the use of low sodium Electrolyte Maintenance Solutions (EMS) has become the standard of care. However, given that North American children infrequently develop severe dehydration, it is unclear if the routine use of EMS is justified. When pediatricians directly dispense EMS, 16 children need to be treated to prevent 1 unscheduled office visit, however the upper bound of the 95% confidence interval is an astounding 508 patients. In addition, EMS is considered by some to be prohibitively expensive, with 15% of pediatricians believing it to be too expensive for their patients to purchase. An additional 40% report that taste is a major barrier to consumption. As a result, oral fluid replenishment is often underutilized and IV rehydration employed instead. Our goal is to provide evidence to guide the selection of the optimal ORT fluids in low-risk children, thus increasing its use, enhancing its success, and reducing the reliance on intravenous rehydration. We hypothesize that the strict adherence to EMS use in low-risk children may actually be counterproductive by resulting in reduced fluid intake and potentially increasing the use of intravenous rehydration.

ELIGIBILITY:
Inclusion Criteria:

* ≥3 episodes of vomiting or diarrhea in preceding 24 hours
* Duration of illness less than 96 hours
* Age 6 - 60 months
* Clinical suspicion of acute intestinal infectious process
* Weight ≥ 8 kg
* Clinical dehydration score < 5
* Capillary refill < 2 seconds
* Absence of bulging fontanelle
* Absence of bilious vomiting
* Absence of blood in diarrhea/emesis
* Absence of abdominal pain (if present reported as periumbilical in location)
* Absence of abdominal distention
* Absence of acute disease currently requiring treatment
* Absence of co-existing diseases (prematurity, cardiac, renal, neurological, metabolic, endocrine, immunodeficiency, trauma or history of ingestion)

Exclusion Criteria:

* Known gastrointestinal diseases (ie. inflammatory bowel disease, celiac) or any other underlying disease process that might place the child at an increased risk of treatment failure.
* Age < 6 months
* Weight < 8 kg
* If premature, corrected gestational age < 30 weeks
* Presence of hematochezia
* Responsible physician judges the child requires immediate intravenous rehydration
* English language is so limited that consent and/or follow-up is not possible.
* Non-Ontario resident [Canadian Institute for Health Information (CIHI) follow-up data will not be available]

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 624 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of children experiencing a treatment failure | Within 7 days of enrolment
  This outcome will be deemed to have occurred if any of the following occur:
  * Requires an unscheduled visit after the initial encounter
  * Requires physician evaluation during a follow-up assessment.
  * Hospitalization or Intravenous Rehydration
  * Extended Symptomatology
  * Failure to consume sufficient study fluid during the initial ED visit

SECONDARY OUTCOMES:
Percent Weight Change | 72-84 hours after enrolment
Proportion of Subjects Receiving Intravenous Rehydration | 7 days
Proportion of Subjects Requiring Hospitalization | 7 days
Frequency of diarrhea and vomiting episodes | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Freedman SB, Willan AR, Boutis K, Schuh S. Effect of Dilute Apple Juice and Preferred Fluids vs Electrolyte Maintenance Solution on Treatment Failure Among Children With Mild Gastroenteritis: A Randomized Clinical Trial. JAMA. 2016 May 10;315(18):1966-74. doi: 10.1001/jama.2016.5352. PMID 27131100